CLINICAL TRIAL: NCT03240978
Title: An Interventional Study for the Effects of Physical Exercise on the Prevention of Prediabetes in Overweight Chinese: Role of Gut Microbiota and Adipokines
Brief Title: Exercise Intervention for the Prevention of Prediabetes in Overweight Chinese
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: UW-15370
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: PreDiabetes; Insulin Sensitivity
MeSH Terms: conditions — Prediabetic State; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity intervention (Experimental): Exercise intervention at 70 to 80% of estimated heart rate maximum for 12 weeks.
  Interventions: Behavioral: exercise intervention
- Moderate intensity intervention (Experimental): Exercise intervention at 50 to 70% of estimated heart rate maximum for 12 weeks.
  Interventions: Behavioral: exercise intervention
- non-exercise group (No Intervention): Participants will not receive any type of exercise training.

INTERVENTIONS:
Behavioral: exercise intervention — A period of 12-week exercise intervention under the supervision of exercise specialists will be conducted.
  Arms: High intensity intervention; Moderate intensity intervention

SUMMARY:
Overweight/obese Chinese and prediabetes will be recruited and divided into three age-matched groups including high intensity exercise, moderate intensity exercise, and non-exercise groups. The exercise program will consist of three sessions per week over the course of 12 weeks, under the supervision of our in-house exercise specialists and physiologists. The effects of exercise on glucose and lipid profiles, insulin sensitivity and adiposity will be evaluated.

DETAILED DESCRIPTION:
60 Chinese men aged between 21 and 60 years old with overweight/obesity (25 kg/m2 <BMI < 32.5 kg/m2) and prediabetes will be recruited.The participants will be divided into three age-matched groups (n=20 in each group),including high intensity exercise, moderate intensity exercise, and non-exercise groups. The suitability of each participant for physical exercise will be assessed by an in-house exercise specialist, based on parameters of blood pressure, strength, cardiovascular fitness, balance, flexibility. The exercise program will consist of three sessions per week over the course of 12 weeks, under the supervision of our in-house exercise specialists and physiologists. Each session will comprise of warm-up, resistance and aerobic training components and a cool-down. The high intensity training (aerobic combined with strength training) will consist of six exercises of three sets each, with each exercise set at an intensity of 6 to 10 repetition maximum. Intensity, volume and exercise selection will be varied both within the week and over the 12 week program in a periodised system designed to maximize muscle hypertrophy and strength gain. Exercise intensity will be at 60 to 80% of estimated heart rate maximum. Moderate intensity training (Aerobic training) will be conducted on a variety of ergometers including treadmill, cycle, rowing and cross training machines. The non-exercise group (delayed group) will be used as placebo control, and will participate in the training group at the later stage.

ELIGIBILITY:
Inclusion Criteria:

- overweight/obese Chinese man (25 kg/m2<BMI<32.5 kg/m2) aged between 21 and 60 years old; prediabetes, impaired glucose tolerance (mean 2-h blood glucose ≥7.8 and ≤11.1 mmol/l after a 75-g oral glucose challenge) or impaired fasting glucose (mean fasting blood glucose ≥6.1 mmol/l and ≤7.0 mmol/l and HbA1c levels between 5.7% and 6.4%).

Exclusion Criteria:

- any neurological, musculoskeletal or cardio respiratory condition, which would put them at risk during exercise or inhibit their ability to adapt to an exercise program; any subject participated in a regular vigorous exercise and/or diet program more than 2 times per week in the 3 months prior to recruitment; any subject who is taking medicine, especially antibiotics in the past week prior to study.

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
change of fasting glucose | change from baseline fasting glucose level at 12 weeks
  fasting glucose level

SECONDARY OUTCOMES:
alterations of gut microbiome | before, 4 weeks and 12 weeks after exercise training
  advanced metagenomics to identify gut microbiota species altered by exercise training
rate of non-responsiveness in the alleviation of insulin resistance to exercise intervention | before and after 12 weeks after exercise training
  Participants in the exercise arms are further classified into responders or non-responsders, depending on whether they could demonstrate a decrease of insulin resistance index (HOMA-IR) greater than 2-fold technical error, which is a threshold for true physiological adaptation. HOMA-IR is calculated using homeostasis model assessment methods, defined as fasting insulin (μU/mL)×fasting glucose (mmol/L)/22.5.

CONTACTS AND LOCATIONS:
Overall Officials: Aimin Xu, Principal Investigator — Department of Medicine, The University of Hong Kong
Locations (1):
- Department of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Chen J, Ni Y, Liu Y, Gao X, Tse MA, Panagiotou G, Xu A. Exercise-changed gut mycobiome as a potential contributor to metabolic benefits in diabetes prevention: an integrative multi-omics study. Gut Microbes. 2024 Jan-Dec;16(1):2416928. doi: 10.1080/19490976.2024.2416928. Epub 2024 Oct 29. PMID 39473051
- [Derived] Jin L, Geng L, Ying L, Shu L, Ye K, Yang R, Liu Y, Wang Y, Cai Y, Jiang X, Wang Q, Yan X, Liao B, Liu J, Duan F, Sweeney G, Woo CWH, Wang Y, Xia Z, Lian Q, Xu A. FGF21-Sirtuin 3 Axis Confers the Protective Effects of Exercise Against Diabetic Cardiomyopathy by Governing Mitochondrial Integrity. Circulation. 2022 Nov 15;146(20):1537-1557. doi: 10.1161/CIRCULATIONAHA.122.059631. Epub 2022 Sep 22. PMID 36134579
- [Derived] Liu Y, Wang Y, Ni Y, Cheung CKY, Lam KSL, Wang Y, Xia Z, Ye D, Guo J, Tse MA, Panagiotou G, Xu A. Gut Microbiome Fermentation Determines the Efficacy of Exercise for Diabetes Prevention. Cell Metab. 2020 Jan 7;31(1):77-91.e5. doi: 10.1016/j.cmet.2019.11.001. Epub 2019 Nov 27. PMID 31786155